CLINICAL TRIAL: NCT05608005
Title: A Parallel-group, Phase I/II, Randomized, Modified Double-blind, 3-arm, Active Comparator, Multi-center, Prevention Study to Evaluate the Immunogenicity and Safety of Two Adjuvanted Dose Levels of Panblok H7+MF59 Influenza Vaccine Compared With an Unadjuvanted Dose of Panblok H7 in Participants 18 Years of Age and Older
Brief Title: Study on Two Adjuvanted Dose Levels of Panblok H7+MF59 Compared for Immunogenicity and Safety With an Unadjuvanted Dose of Panblok H7 in Participants 18 Years of Age and Older
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: VAM00001; U1111-1256-9115 (Registry Identifier: ICTRP)
Expanded Access: Available
Record Dates: First submitted 2022-10-20; First posted 2022-11-07 (Actual); Results first posted 2025-02-20 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Influenza; Healthy Volunteers
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Intervention Model Description: Eligible participants (18-64 years of age and ≥65 years of age) will be randomized in a 3:3:1 ratio to receive 2 doses, 21 days apart, by intramuscular (IM) route of either Panblok H7+MF59 (dose 1), Panblok H7+MF59 (dose 2), or unadjuvanted Panblok H7 (dose 3) at D01.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Modified double-blind:
  * Investigators and study staff who conduct the safety assessment, laboratory personnel who analyze the blood samples, Sponsor's personnel and study Team members, and the participant will not know which study dose is administered
  * Only the study staff who prepare and administer the study intervention and are not involved with the safety evaluation will know which study dose is administered
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group 1 (Experimental): 2 doses, 21 days apart, of Panblok H7 dose 1 + MF59
  Interventions: Biological: Panblok + MF59 Dose 1
- Group 2 (Experimental): 2 doses, 21 days apart, of Panblok H7 dose 2 + MF59
  Interventions: Biological: Panblok + MF59 Dose 2
- Group 3 (Active Comparator): 2 doses, 21 days apart, of Panblok H7 dose 3 unadjuvanted
  Interventions: Biological: Unadjuvanted Panblok Dose 3

INTERVENTIONS:
Biological: Panblok + MF59 Dose 1 — Pharmaceutical form: suspension for injection Route of administration: intramuscular
  Arms: Group 1
Biological: Panblok + MF59 Dose 2 — Pharmaceutical form: suspension for injection Route of administration: intramuscular
  Arms: Group 2
Biological: Unadjuvanted Panblok Dose 3 — Pharmaceutical form: liquid for injection Route of administration: intramuscular
  Arms: Group 3

SUMMARY:
VAM00001 is a Phase I/II, randomized, modified double-blind, multi-center study.

The purpose of this study is to compare 2 dose levels of Panblok H7 (dose 1 and dose 2 of rHA) with a standard squalene dose of adjuvant MF59 to Panblok H7 (dose 3) unadjuvanted in approximately 700 adult participants in order to select one dose formulation to be used for further clinical development. The randomization ratio will be 3:3:1 for Panblok H7 (dose 1) + MF59, Panblok H7 (dose 2) + MF59, and Panblok H7 (dose 3) unadjuvanted, respectively. Each study group will be stratified into the age groups 18-64 years and ≥ 65 years of age.

The study duration for each participant will be approximately 13 months.

DETAILED DESCRIPTION:
The study duration for each participant will be approximately 13 months.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older on the day of inclusion
* Participants who are healthy as determined by medical evaluation including medical history and physical examination
* A female participant is eligible to participate if she is not pregnant or breastfeeding and one of the following conditions applies:

Is of non-childbearing potential. To be considered of non-childbearing potential, a female must be post-menopausal for at least 1 year, or surgically sterile.

OR Is of childbearing potential and agrees to use a highly effective contraceptive method or abstinence from at least 4 weeks prior to each study intervention administration until at least 12 weeks after the last study intervention administration.

* A female participant of childbearing potential must have a negative highly sensitive pregnancy test (urine or serum as required by local regulation) within 24 hours before the first dose of study intervention
* Informed consent form has been signed and dated

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy, within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months)
* Known systemic hypersensitivity to any of the study intervention components, or history of a life-threatening reaction to the study interventions used in the study or to a product containing any of the same substances
* Thrombocytopenia or bleeding disorder contraindicating intramuscular injection based on investigator's judgement
* Chronic illness that, in the opinion of the investigator, is at a stage where it might interfere with study conduct or completion (1)

  (1) Chronic illness may include, but is not limited to, cardiac disorders, renal disorders, auto-immune disorders, diabetes, psychiatric disorders, or chronic infection
* Neoplastic disease or any hematologic malignancy (except localized skin or prostate cancer that is stable at the time of study intervention administration in the absence of therapy, and participants who have a history of neoplastic disease and who have been disease-free for ≥ 5 years)
* Moderate or severe acute illness/infection (according to investigator judgment) or febrile illness (temperature ≥ 100.4°F) on the day of study intervention administration. A prospective participant should not be included in the study until the condition has resolved or the febrile event has subsided
* Alcohol, prescription drug, or substance abuse that, in the opinion of the Investigator, might interfere with the study conduct or completion
* Receipt of any vaccine in the 14 days preceding Visit 1 or planned receipt of any vaccine prior to Visit 3, except for seasonal flu vaccine, which may be received at least 2 weeks after Visit 2
* Previous vaccination against H7N9 with an investigational vaccine
* Receipt of immune globulins, blood or blood-derived products in the past 3 months
* Participation at the time of study enrollment (or in the 4 weeks preceding the first study intervention administration) or planned participation during the present study period in another clinical study investigating a vaccine, drug, medical device, or medical procedure
* Deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized involuntarily
* Identified as an Investigator or employee of the Investigator or study center with direct involvement in the proposed study, or identified as an immediate family member (ie, parent, spouse, natural or adopted child) of the Investigator or employee with direct involvement in the proposed study
* Personal or family history of Guillain-Barré syndrome
* Self-reported seropositivity for Hepatitis B antigen or Hepatitis C

"The above information is not intended to contain all considerations relevant to a potential participation in a clinical trial."

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 581 (Actual)
Dates: Start 2022-11-03 (Actual); Primary Completion 2023-02-18 (Actual); Study Completion 2024-02-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — MCM Vaccines B.V.
Locations (16):
- United States (16):
  - Centricity Research-Mesa Site Number : 8400006, Mesa, Arizona
  - Velocity Clinical Research-Hallandale Beach Site Number : 8400026, Hallandale, Florida
  - Research Centers of America Site Number : 8400024, Hollywood, Florida
  - Suncoast Research Associates, LLC Site Number : 8400008, Miami, Florida
  - St Johns Center for Clinical Research Site Number : 8400021, Saint Augustine, Florida
  - CenExel ACMR (Atlanta Center for Medical Research) Site Number : 8400022, Atlanta, Georgia
  - Velocity Clinical Research Valparaiso Site Number : 8400007, Valparaiso, Indiana
  - Velocity Clinical Research Site Number : 8400027, Metairie, Louisiana
  - M3 Wake Research Inc Site Number : 8400010, Raleigh, North Carolina
  - Preferred Primary Care Physicians Site Number : 8400015, Pittsburgh, Pennsylvania
  - Preferred Primary Care Physicians, Inc. Site Number : 8400002, Pittsburgh, Pennsylvania
  - Velocity Clinical Research Anderson Site Number : 8400016, Anderson, South Carolina
  - WR-ClinSearch, LLC Site Number : 8400003, Chattanooga, Tennessee
  - Velocity Clinical Research Site Number : 8400019, Austin, Texas
  - JBR Clinical Research Site Number : 8400005, Salt Lake City, Utah
  - Foothill Family Research-South Site Number : 8400009, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: VAM00001 Plain Language Results Summary — https://sanofi.trialsummaries.com/Study/StudyDetails?id=25367&tenant=MT_SNY_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 16 centers in the United States between 03 November 2022 and 13 February 2024.
Pre-assignment Details: A total of 581 participants were enrolled and randomized in the study.
Groups:
- Group 1: Panblok H7 (7.5 mcg) + MF59: Participants received panblok H7 7.5 microgram (mcg) + MF59 adjuvant intramuscular (IM) injection once daily on Days 1 and 22.
- Group 2: Panblok H7 (15 mcg) + MF59: Participants received panblok H7 15 mcg + MF59 adjuvant IM injection once daily on Days 1 and 22.
- Group 3: Panblok H7 (45 mcg) Unadjuvanted: Participants received panblok H7 45 mcg unadjuvanted IM injection once daily on Days 1 and 22.
Period: Overall Study
Arm/Group | Group 1: Panblok H7 (7.5 mcg) + MF59 | Group 2: Panblok H7 (15 mcg) + MF59 | Group 3: Panblok H7 (45 mcg) Unadjuvanted
Started | 248 | 249 | 84
Vaccinated | 243 | 246 | 84
Completed | 203 | 199 | 62
Not Completed | 45 | 50 | 22
Not completed — Adverse Event | 2 | 1 | 3
Not completed — Protocol Violation | 2 | 3 | 0
Not completed — Withdrawal by Subject | 10 | 12 | 4
Not completed — Lost to Follow-up | 25 | 27 | 15
Not completed — Participants were not vaccinated or withdrew for other reasons | 6 | 7 | 0

BASELINE CHARACTERISTICS:
Population: The Safety analysis set included all participants who had received at least 1 study vaccine.
Groups:
- Group 1: Panblok H7 (7.5 mcg) + MF59: Participants received panblok H7 7.5 mcg + MF59 adjuvant IM injection once daily on Days 1 and 22.
- Total: Total of all reporting groups
Arm/Group | Group 1: Panblok H7 (7.5 mcg) + MF59 | Group 2: Panblok H7 (15 mcg) + MF59 | Group 3: Panblok H7 (45 mcg) Unadjuvanted | Total
Number analyzed (Participants) | 243 | 246 | 84 | 573
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.6 (15.2) | 56.2 (15.3) | 54.7 (17.1) | 56.2 (15.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 127 | 125 | 47 | 299
  Male | 116 | 121 | 37 | 274
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 0 | 3
  Asian | 1 | 1 | 0 | 2
  Black or African American | 67 | 62 | 17 | 146
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 0 | 2
  White | 168 | 173 | 67 | 408
  Multiple origin | 0 | 2 | 0 | 2
  Not Reported | 4 | 2 | 0 | 6
  Unknown | 1 | 3 | 0 | 4

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean of Hemagglutination Inhibition (HAI) Antibody (Ab) Titer at Day 22
Description: The HAI antibody was measured by hemagglutination inhibition using horse red blood cells (HIH) measurement method. The 95% confidence interval (CI) was based on the Student t-distribution of log10-transformed values.
Time Frame: Day 22
Population: The Full analysis set (FAS) included all randomized participants who received at least 1 dose of the study vaccine and had a post-vaccination blood sample for Day 22 or Day 43. Only participants analyzed at Day 22 are reported.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Group 1: Panblok H7 (7.5 mcg) + MF59 | Group 2: Panblok H7 (15 mcg) + MF59 | Group 3: Panblok H7 (45 mcg) Unadjuvanted
Number analyzed (Participants) | 231 | 232 | 76
titer | 5.74 [5.44 to 6.06] | 5.61 [5.34 to 5.90] | 5.28 [5.10 to 5.47]

2. Primary Outcome: Geometric Mean of Hemagglutination Inhibition Antibody Titer at Day 43
Description: The HAI antibody was measured by HIH measurement method. The 95% CI was based on the Student t-distribution of log10-transformed values.
Time Frame: Day 43
Population: The FAS included all randomized participants who received at least 1 dose of the study vaccine and had a post-vaccination blood sample for Day 22 or Day 43. Only participants analyzed at Day 43 are reported.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Group 1: Panblok H7 (7.5 mcg) + MF59 | Group 2: Panblok H7 (15 mcg) + MF59 | Group 3: Panblok H7 (45 mcg) Unadjuvanted
Number analyzed (Participants) | 224 | 231 | 72
titer | 12.6 [10.8 to 14.6] | 13.4 [11.6 to 15.5] | 5.80 [5.37 to 6.27]

3. Primary Outcome: Geometric Mean Ratio of Hemagglutination Inhibition Antibody Titer at Day 22
Description: The HAI antibody was measured by HIH measurement method. The geometric mean ratio of antibody titer at post-vaccination over pre-vaccination is reported. The 95% CI was based on the Student t-distribution of log10-transformed values.
Time Frame: Days 1 and 22
Population: The FAS included all randomized participants who received at least 1 dose of the study vaccine and had a post-vaccination blood sample for Day 22 or Day 43. Only participants analyzed at Days 1 and 22 are reported.
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Group 1: Panblok H7 (7.5 mcg) + MF59 | Group 2: Panblok H7 (15 mcg) + MF59 | Group 3: Panblok H7 (45 mcg) Unadjuvanted
Number analyzed (Participants) | 230 | 232 | 76
ratio | 1.09 [1.03 to 1.15] | 1.05 [0.998 to 1.11] | 1.03 [0.981 to 1.08]

4. Primary Outcome: Geometric Mean Ratio of Hemagglutination Inhibition Antibody Titer at Day 43
Description: as for outcome 3
Time Frame: Days 1 and 43
Population: The FAS included all randomized participants who received at least 1 dose of the study vaccine and had a post-vaccination blood sample for Day 22 or Day 43. Only participants analyzed at Days 1 and 43 are reported.
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Group 1: Panblok H7 (7.5 mcg) + MF59 | Group 2: Panblok H7 (15 mcg) + MF59 | Group 3: Panblok H7 (45 mcg) Unadjuvanted
Number analyzed (Participants) | 223 | 231 | 72
ratio | 2.39 [2.05 to 2.78] | 2.52 [2.17 to 2.91] | 1.13 [1.05 to 1.23]

5. Primary Outcome: Geometric Mean Ratio of Hemagglutination Inhibition Antibody Titer at Day 202
Description: as for outcome 3
Time Frame: Days 1 and 202
Population: The FAS included all randomized participants who received at least 1 dose of the study vaccine and had a post-vaccination blood sample for Day 22 or Day 43. Only participants analyzed at Days 1 and 202 are reported.
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Group 1: Panblok H7 (7.5 mcg) + MF59 | Group 2: Panblok H7 (15 mcg) + MF59 | Group 3: Panblok H7 (45 mcg) Unadjuvanted
Number analyzed (Participants) | 209 | 212 | 66
ratio | 1.01 [0.969 to 1.05] | 0.966 [0.920 to 1.01] | 0.990 [0.951 to 1.03]

6. Primary Outcome: Geometric Mean Ratio of Hemagglutination Inhibition Antibody Titer at Day 387
Description: as for outcome 3
Time Frame: Days 1 and 387
Population: The FAS included all randomized participants who received at least 1 dose of the study vaccine and had a post-vaccination blood sample for Day 22 or Day 43. Only participants analyzed at Days 1 and 387 are reported.
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Group 1: Panblok H7 (7.5 mcg) + MF59 | Group 2: Panblok H7 (15 mcg) + MF59 | Group 3: Panblok H7 (45 mcg) Unadjuvanted
Number analyzed (Participants) | 202 | 198 | 61
ratio | 0.998 [0.961 to 1.04] | 0.976 [0.927 to 1.03] | 0.978 [0.943 to 1.01]

7. Primary Outcome: Percentage of Participants With Seroconversion of Hemagglutination Inhibition Antibody Titer at Day 22
Description: The seroconversion was defined as titer <10 on Day 1 and post-injection titer >=40 on Day 22 or Day 43; or defined as titer >=10 on Day 1 and a >=4-fold increase in titer on Day 22 or Day 43. The 95% CI for the single percentage was based on the Clopper-Pearson method. The percentages are rounded off to the tenth decimal place.
Time Frame: Day 22
Population: The FAS included all randomized participants who received at least 1 dose of the study vaccine and had a post-vaccination blood sample for Day 22 or Day 43. Only participants analyzed at Day 22 are reported.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: Panblok H7 (7.5 mcg) + MF59 | Group 2: Panblok H7 (15 mcg) + MF59 | Group 3: Panblok H7 (45 mcg) Unadjuvanted
Number analyzed (Participants) | 230 | 232 | 76
percentage of participants | 2.2 [0.7 to 5.0] | 0.4 [0.0 to 2.4] | 0.0 [0.0 to 4.7]

8. Primary Outcome: Percentage of Participants With Seroconversion of Hemagglutination Inhibition Antibody Titer at Day 43
Description: as for outcome 7
Time Frame: Day 43
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: Panblok H7 (7.5 mcg) + MF59 | Group 2: Panblok H7 (15 mcg) + MF59 | Group 3: Panblok H7 (45 mcg) Unadjuvanted
Number analyzed (Participants) | 223 | 231 | 72
percentage of participants | 22.9 [17.5 to 28.9] | 22.9 [17.7 to 28.9] | 1.4 [0.0 to 7.5]

9. Primary Outcome: Percentage of Participants With Hemagglutination Inhibition Antibody Titer >=1:40 at Day 1
Description: The HAI antibody was measured by HIH measurement method. The 95% CI for the single percentage was based on the Clopper-Pearson method. The percentages are rounded off to the tenth decimal place.
Time Frame: Day 1
Population: The FAS included all randomized participants who received at least 1 dose of the study vaccine and had a post-vaccination blood sample for Day 22 or Day 43. Only participants analyzed at Day 1 are reported.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: Panblok H7 (7.5 mcg) + MF59 | Group 2: Panblok H7 (15 mcg) + MF59 | Group 3: Panblok H7 (45 mcg) Unadjuvanted
Number analyzed (Participants) | 233 | 233 | 76
percentage of participants | 0.0 [0.0 to 1.6] | 0.9 [0.1 to 3.1] | 0.0 [0.0 to 4.7]

10. Primary Outcome: Percentage of Participants With Hemagglutination Inhibition Antibody Titer >=1:40 at Day 22
Description: as for outcome 9
Time Frame: Day 22
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: Panblok H7 (7.5 mcg) + MF59 | Group 2: Panblok H7 (15 mcg) + MF59 | Group 3: Panblok H7 (45 mcg) Unadjuvanted
Number analyzed (Participants) | 231 | 232 | 76
percentage of participants | 2.2 [0.7 to 5.0] | 0.9 [0.1 to 3.1] | 0.0 [0.0 to 4.7]

11. Primary Outcome: Percentage of Participants With Hemagglutination Inhibition Antibody Titer >=1:40 at Day 43
Description: as for outcome 9
Time Frame: Day 43
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: Panblok H7 (7.5 mcg) + MF59 | Group 2: Panblok H7 (15 mcg) + MF59 | Group 3: Panblok H7 (45 mcg) Unadjuvanted
Number analyzed (Participants) | 224 | 231 | 72
percentage of participants | 23.2 [17.9 to 29.3] | 23.4 [18.1 to 29.4] | 1.4 [0.0 to 7.5]

12. Primary Outcome: Percentage of Participants With Hemagglutination Inhibition Antibody Titer >=1:40 at Day 202
Description: as for outcome 9
Time Frame: Day 202
Population: The FAS included all randomized participants who received at least 1 dose of the study vaccine and had a post-vaccination blood sample for Day 22 or Day 43. Only participants analyzed at Day 202 are reported.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: Panblok H7 (7.5 mcg) + MF59 | Group 2: Panblok H7 (15 mcg) + MF59 | Group 3: Panblok H7 (45 mcg) Unadjuvanted
Number analyzed (Participants) | 210 | 212 | 66
percentage of participants | 0.5 [0.0 to 2.6] | 0.0 [0.0 to 1.7] | 0.0 [0.0 to 5.4]

13. Primary Outcome: Percentage of Participants With Hemagglutination Inhibition Antibody Titer >=1:40 at Day 387
Description: as for outcome 9
Time Frame: Day 387
Population: The FAS included all randomized participants who received at least 1 dose of the study vaccine and had a post-vaccination blood sample for Day 22 or Day 43. Only participants analyzed at Day 387 are reported.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: Panblok H7 (7.5 mcg) + MF59 | Group 2: Panblok H7 (15 mcg) + MF59 | Group 3: Panblok H7 (45 mcg) Unadjuvanted
Number analyzed (Participants) | 203 | 198 | 61
percentage of participants | 0.0 [0.0 to 1.8] | 0.0 [0.0 to 1.8] | 0.0 [0.0 to 5.9]

14. Primary Outcome: Percentage of Participants With Detectable Hemagglutination Inhibition Antibody Titer >=1:10 at Day 1
Description: as for outcome 9
Time Frame: Day 1
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: Panblok H7 (7.5 mcg) + MF59 | Group 2: Panblok H7 (15 mcg) + MF59 | Group 3: Panblok H7 (45 mcg) Unadjuvanted
Number analyzed (Participants) | 233 | 233 | 76
percentage of participants | 3.4 [1.5 to 6.7] | 3.4 [1.5 to 6.7] | 1.3 [0.0 to 7.1]

15. Primary Outcome: Percentage of Participants With Detectable Hemagglutination Inhibition Antibody Titer >=1:10 at Day 22
Description: as for outcome 9
Time Frame: Day 22
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: Panblok H7 (7.5 mcg) + MF59 | Group 2: Panblok H7 (15 mcg) + MF59 | Group 3: Panblok H7 (45 mcg) Unadjuvanted
Number analyzed (Participants) | 231 | 232 | 76
percentage of participants | 6.9 [4.0 to 11.0] | 6.5 [3.7 to 10.4] | 2.6 [0.3 to 9.2]

16. Primary Outcome: Percentage of Participants With Detectable Hemagglutination Inhibition Antibody Titer >=1:10 at Day 43
Description: as for outcome 9
Time Frame: Day 43
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: Panblok H7 (7.5 mcg) + MF59 | Group 2: Panblok H7 (15 mcg) + MF59 | Group 3: Panblok H7 (45 mcg) Unadjuvanted
Number analyzed (Participants) | 224 | 231 | 72
percentage of participants | 46.9 [40.2 to 53.6] | 52.4 [45.7 to 59.0] | 9.7 [4.0 to 19.0]

17. Primary Outcome: Percentage of Participants With Detectable Hemagglutination Inhibition Antibody Titer >=1:10 at Day 202
Description: as for outcome 9
Time Frame: Day 202
Population: as for outcome 12
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: Panblok H7 (7.5 mcg) + MF59 | Group 2: Panblok H7 (15 mcg) + MF59 | Group 3: Panblok H7 (45 mcg) Unadjuvanted
Number analyzed (Participants) | 210 | 212 | 66
percentage of participants | 3.3 [1.4 to 6.7] | 2.4 [0.8 to 5.4] | 1.5 [0.0 to 8.2]

18. Primary Outcome: Percentage of Participants With Detectable Hemagglutination Inhibition Antibody Titer >=1:10 at Day 387
Description: as for outcome 9
Time Frame: Day 387
Population: as for outcome 13
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: Panblok H7 (7.5 mcg) + MF59 | Group 2: Panblok H7 (15 mcg) + MF59 | Group 3: Panblok H7 (45 mcg) Unadjuvanted
Number analyzed (Participants) | 203 | 198 | 61
percentage of participants | 3.0 [1.1 to 6.3] | 2.5 [0.8 to 5.8] | 0.0 [0.0 to 5.9]

19. Primary Outcome: Geometric Mean of Neutralization Test (NT) Antibody Titer at Day 22
Description: The NT antibody was measured by seroneutralization (SN) measurement method. The 95% CI was based on the Student t-distribution of log10-transformed values.
Time Frame: Day 22
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Group 1: Panblok H7 (7.5 mcg) + MF59 | Group 2: Panblok H7 (15 mcg) + MF59 | Group 3: Panblok H7 (45 mcg) Unadjuvanted
Number analyzed (Participants) | 231 | 232 | 76
titer | 7.23 [6.61 to 7.91] | 6.85 [6.31 to 7.45] | 6.88 [6.04 to 7.84]

20. Primary Outcome: Geometric Mean of Neutralization Test Antibody Titer at Day 43
Description: The NT antibody was measured by SN measurement method. The 95% CI was based on the Student t-distribution of log10-transformed values.
Time Frame: Day 43
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Group 1: Panblok H7 (7.5 mcg) + MF59 | Group 2: Panblok H7 (15 mcg) + MF59 | Group 3: Panblok H7 (45 mcg) Unadjuvanted
Number analyzed (Participants) | 224 | 231 | 72
titer | 26.8 [22.0 to 32.6] | 25.8 [21.9 to 30.4] | 11.5 [9.31 to 14.1]

21. Primary Outcome: Geometric Mean Ratio of Neutralization Test Antibody Titer at Day 22
Description: The NT antibody was measured by SN measurement method. The geometric mean ratio of antibody titer at post-vaccination over pre-vaccination is reported. The 95% CI was based on the Student t-distribution of log10-transformed values.
Time Frame: Days 1 and 22
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Group 1: Panblok H7 (7.5 mcg) + MF59 | Group 2: Panblok H7 (15 mcg) + MF59 | Group 3: Panblok H7 (45 mcg) Unadjuvanted
Number analyzed (Participants) | 230 | 232 | 76
ratio | 1.21 [1.09 to 1.35] | 1.14 [1.04 to 1.25] | 1.09 [0.923 to 1.28]

22. Primary Outcome: Geometric Mean Ratio of Neutralization Test Antibody Titer at Day 43
Description: as for outcome 21
Time Frame: Days 1 and 43
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Group 1: Panblok H7 (7.5 mcg) + MF59 | Group 2: Panblok H7 (15 mcg) + MF59 | Group 3: Panblok H7 (45 mcg) Unadjuvanted
Number analyzed (Participants) | 223 | 231 | 72
ratio | 4.51 [3.66 to 5.55] | 4.29 [3.59 to 5.14] | 1.86 [1.46 to 2.38]

23. Primary Outcome: Geometric Mean Ratio of Neutralization Test Antibody Titer at Day 202
Description: as for outcome 21
Time Frame: Days 1 and 202
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Group 1: Panblok H7 (7.5 mcg) + MF59 | Group 2: Panblok H7 (15 mcg) + MF59 | Group 3: Panblok H7 (45 mcg) Unadjuvanted
Number analyzed (Participants) | 209 | 212 | 66
ratio | 1.20 [1.07 to 1.34] | 1.17 [1.05 to 1.30] | 0.856 [0.735 to 0.997]

24. Primary Outcome: Geometric Mean Ratio of Neutralization Test Antibody Titer at Day 387
Description: as for outcome 21
Time Frame: Days 1 and 387
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Group 1: Panblok H7 (7.5 mcg) + MF59 | Group 2: Panblok H7 (15 mcg) + MF59 | Group 3: Panblok H7 (45 mcg) Unadjuvanted
Number analyzed (Participants) | 202 | 198 | 61
ratio | 1.20 [1.07 to 1.35] | 1.18 [1.06 to 1.32] | 0.909 [0.792 to 1.04]

25. Primary Outcome: Percentage of Participants With Neutralization Test Antibody Titer >=1:20, >=1:40, and >=1:80 at Day 22
Description: The NT antibody was measured by SN measurement method. The 95% CI was the single percentage was based on the Clopper-Pearson method. The percentages are rounded off to the tenth decimal place.
Time Frame: Day 22
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: Panblok H7 (7.5 mcg) + MF59 | Group 2: Panblok H7 (15 mcg) + MF59 | Group 3: Panblok H7 (45 mcg) Unadjuvanted
Number analyzed (Participants) | 231 | 232 | 76
percentage of participants
  Antibody Titer >=1:20 | 10.0 [6.4 to 14.6] | 7.3 [4.3 to 11.5] | 7.9 [3.0 to 16.4]
  Antibody Titer >=1:40 | 2.2 [0.7 to 5.0] | 2.2 [0.7 to 5.0] | 0.0 [0.0 to 4.7]
  Antibody Titer >=1:80 | 1.3 [0.3 to 3.7] | 0.9 [0.1 to 3.1] | 0.0 [0.0 to 4.7]

26. Primary Outcome: Percentage of Participants With Neutralization Test Antibody Titer >=1:20, >=1:40, and >=1:80 at Day 43
Description: as for outcome 25
Time Frame: Day 43
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: Panblok H7 (7.5 mcg) + MF59 | Group 2: Panblok H7 (15 mcg) + MF59 | Group 3: Panblok H7 (45 mcg) Unadjuvanted
Number analyzed (Participants) | 224 | 231 | 72
percentage of participants
  Antibody Titer >=1:20 | 54.9 [48.1 to 61.5] | 55.8 [49.2 to 62.4] | 29.2 [19.0 to 41.1]
  Antibody Titer >=1:40 | 35.7 [29.4 to 42.4] | 35.1 [28.9 to 41.6] | 11.1 [4.9 to 20.7]
  Antibody Titer >=1:80 | 22.3 [17.0 to 28.3] | 16.0 [11.5 to 21.4] | 2.8 [0.3 to 9.7]

27. Primary Outcome: Percentage of Participants With >=2 and >=4 Fold Increase in Neutralization Test Antibody Titer at Day 22
Description: as for outcome 25
Time Frame: Day 22
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: Panblok H7 (7.5 mcg) + MF59 | Group 2: Panblok H7 (15 mcg) + MF59 | Group 3: Panblok H7 (45 mcg) Unadjuvanted
Number analyzed (Participants) | 230 | 232 | 76
percentage of participants
  >=2 fold increase | 22.2 [17.0 to 28.1] | 17.2 [12.6 to 22.7] | 18.4 [10.5 to 29.0]
  >=4 fold increase | 7.8 [4.7 to 12.1] | 6.0 [3.3 to 9.9] | 5.3 [1.5 to 12.9]

28. Primary Outcome: Percentage of Participants With >=2 and >=4 Fold Increase in Neutralization Test Antibody Titer at Day 43
Description: as for outcome 25
Time Frame: Day 43
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: Panblok H7 (7.5 mcg) + MF59 | Group 2: Panblok H7 (15 mcg) + MF59 | Group 3: Panblok H7 (45 mcg) Unadjuvanted
Number analyzed (Participants) | 223 | 231 | 72
percentage of participants
  >=2 fold increase | 64.6 [57.9 to 70.8] | 71.4 [65.1 to 77.2] | 48.6 [36.7 to 60.7]
  >=4 fold increase | 51.1 [44.4 to 57.9] | 51.9 [45.3 to 58.5] | 26.4 [16.7 to 38.1]

29. Primary Outcome: Percentage of Participants With Detectable Neutralization Test Antibody Titer >=1:10 at Day 1
Description: as for outcome 25
Time Frame: Day 1
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: Panblok H7 (7.5 mcg) + MF59 | Group 2: Panblok H7 (15 mcg) + MF59 | Group 3: Panblok H7 (45 mcg) Unadjuvanted
Number analyzed (Participants) | 233 | 233 | 76
percentage of participants | 14.2 [10.0 to 19.3] | 15.5 [11.1 to 20.7] | 18.4 [10.5 to 29.0]

30. Primary Outcome: Percentage of Participants With Detectable Neutralization Test Antibody Titer >=1:10 at Day 22
Description: as for outcome 25
Time Frame: Day 22
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: Panblok H7 (7.5 mcg) + MF59 | Group 2: Panblok H7 (15 mcg) + MF59 | Group 3: Panblok H7 (45 mcg) Unadjuvanted
Number analyzed (Participants) | 231 | 232 | 76
percentage of participants | 26.8 [21.2 to 33.0] | 24.1 [18.8 to 30.2] | 26.3 [16.9 to 37.7]

31. Primary Outcome: Percentage of Participants With Detectable Neutralization Test Antibody Titer >=1:10 at Day 43
Description: as for outcome 25
Time Frame: Day 43
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: Panblok H7 (7.5 mcg) + MF59 | Group 2: Panblok H7 (15 mcg) + MF59 | Group 3: Panblok H7 (45 mcg) Unadjuvanted
Number analyzed (Participants) | 224 | 231 | 72
percentage of participants | 69.6 [63.2 to 75.6] | 76.2 [70.2 to 81.5] | 54.2 [42.0 to 66.0]

32. Primary Outcome: Percentage of Participants With Detectable Neutralization Test Antibody Titer >=1:10 at Day 202
Description: as for outcome 25
Time Frame: Day 202
Population: as for outcome 12
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: Panblok H7 (7.5 mcg) + MF59 | Group 2: Panblok H7 (15 mcg) + MF59 | Group 3: Panblok H7 (45 mcg) Unadjuvanted
Number analyzed (Participants) | 210 | 212 | 66
percentage of participants | 25.7 [19.9 to 32.2] | 25.0 [19.3 to 31.4] | 6.1 [1.7 to 14.8]

33. Primary Outcome: Percentage of Participants With Detectable Neutralization Test Antibody Titer >=1:10 at Day 387
Description: as for outcome 25
Time Frame: Day 387
Population: as for outcome 13
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: Panblok H7 (7.5 mcg) + MF59 | Group 2: Panblok H7 (15 mcg) + MF59 | Group 3: Panblok H7 (45 mcg) Unadjuvanted
Number analyzed (Participants) | 203 | 198 | 61
percentage of participants | 24.1 [18.4 to 30.6] | 26.3 [20.3 to 33.0] | 8.2 [2.7 to 18.1]

34. Secondary Outcome: Number of Participants With Immediate Unsolicited Systemic Adverse Events (AEs)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study vaccine, whether or not considered related to the study vaccine. An unsolicited AE is an observed AE that does not fulfill the conditions of solicited reactions, that is, pre-listed in the case report form in terms of diagnosis and onset window post-vaccination. Systemic AEs are all AEs that were not injection or administration site reactions. Immediate events are recorded to capture medically relevant unsolicited systemic AEs which occur within the first 30 minutes after vaccination.
Time Frame: Up to 30 minutes after each vaccination
Population: The Safety analysis set included all participants who had received at least 1 study vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Panblok H7 (7.5 mcg) + MF59 | Group 2: Panblok H7 (15 mcg) + MF59 | Group 3: Panblok H7 (45 mcg) Unadjuvanted
Number analyzed (Participants) | 243 | 246 | 84
Participants | 1 | 0 | 0

35. Secondary Outcome: Number of Participants With Solicited Injection Site Reactions and Systemic Reactions
Description: An adverse reaction (AR) is any noxious and unintended response to a study vaccine related to any dose. A solicited reaction is an "expected" AR (sign or symptom) observed and reported under the conditions (nature and onset) pre-listed in the protocol and case report form. An injection/administration site reaction is an AR at and around the injection/administration site of the investigational medical product. Systemic ARs are all ARs that are not injection or administration site reactions.
Time Frame: Up to 7 days after each vaccination
Population: The Safety analysis set included all participants who had received at least 1 study vaccine. Only participants analyzed for specific parameter are reported.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Panblok H7 (7.5 mcg) + MF59 | Group 2: Panblok H7 (15 mcg) + MF59 | Group 3: Panblok H7 (45 mcg) Unadjuvanted
Number analyzed (Participants) | 242 | 244 | 83
Participants
  Solicited injection site reaction | 53 | 57 | 8
  Solicited systemic reaction: number analyzed (Participants) | 242 | 243 | 83
  Solicited systemic reaction | 57 | 56 | 20

36. Secondary Outcome: Number of Participants With Unsolicited AEs
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study vaccine, whether or not considered related to the study vaccine. An unsolicited AE is an observed AE that does not fulfill the conditions of solicited reactions, that is, pre-listed in the case report form in terms of diagnosis and onset window post-vaccination.
Time Frame: Up to 21 days after each vaccination
Population: The Safety analysis set included all participants who had received at least 1 study vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Panblok H7 (7.5 mcg) + MF59 | Group 2: Panblok H7 (15 mcg) + MF59 | Group 3: Panblok H7 (45 mcg) Unadjuvanted
Number analyzed (Participants) | 243 | 246 | 84
Participants | 32 | 39 | 9

37. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs), Adverse Event of Special Interest (AESIs) and Medically Attended Adverse Events (MAAEs)
Description: An SAE is any untoward medical occurrence that at any dose results in death or is life-threatening or requires inpatient hospitalization or prolongation of existing hospitalization or results in persistent or significant disability/incapacity or is a congenital anomaly/birth defect or is an important medical event. An AESI (serious or non-serious) is one of scientific and medical concern specific to the Sponsor's study vaccine or program, for which ongoing monitoring and rapid communication by the investigator to the Sponsor can be appropriate. An MAAE is a new onset or a worsening of a condition that prompts the participant to seek unplanned medical advice at a physician's office or Emergency Department.
Time Frame: From first dose vaccine administration (Day 1) until 12 months after the last dose administration, 387 days
Population: The Safety analysis set included all participants who had received at least 1 study vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Panblok H7 (7.5 mcg) + MF59 | Group 2: Panblok H7 (15 mcg) + MF59 | Group 3: Panblok H7 (45 mcg) Unadjuvanted
Number analyzed (Participants) | 243 | 246 | 84
Participants
  Any SAE | 11 | 12 | 6
  Any AESI | 1 | 1 | 0
  Any MAAE | 41 | 42 | 10

ADVERSE EVENTS:
Time Frame: From first dose vaccine administration (Day 1) up to 12 months after the last dose administration, maximum of 387 days
Description: The Safety analysis set included all participants who had received at least 1 study vaccine.
Arm/Group | Group 1: Panblok H7 (7.5 mcg) + MF59 | Group 2: Panblok H7 (15 mcg) + MF59 | Group 3: Panblok H7 (45 mcg) Unadjuvanted
All-Cause Mortality (participants affected / at risk) | 1/243 | 1/246 | 0/84
Serious Adverse Events (participants affected / at risk) | 11/243 | 12/246 | 6/84
Other Adverse Events (participants affected / at risk) | 82/243 | 82/246 | 23/84
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: Panblok H7 (7.5 mcg) + MF59 (N=243) | Group 2: Panblok H7 (15 mcg) + MF59 (N=246) | Group 3: Panblok H7 (45 mcg) Unadjuvanted (N=84)
Arteriosclerosis Coronary Artery (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Atrial Flutter (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Coronary Artery Disease (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1)
Mitral Valve Incompetence (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Stress Cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Inguinal Hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Intestinal Obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Small Intestinal Obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Death (General disorders) | 0 (0) | 1 (1) | 0 (0)
Oedema (General disorders) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Clostridium Difficile Infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Fournier's Gangrene (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Pneumonia Respiratory Syncytial Viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Postoperative Wound Infection (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
Salmonellosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Ankle Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Bone Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Fractured Coccyx (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Road Traffic Accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Thermal Burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Traumatic Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Cardiac Myxoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Cardiac Valve Fibroelastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Fallopian Tube Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Lung Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Renal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular Accident (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Embolic Cerebral Infarction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Acute Kidney Injury (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Giant Cell Arteritis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: Panblok H7 (7.5 mcg) + MF59 (N=243) | Group 2: Panblok H7 (15 mcg) + MF59 (N=246) | Group 3: Panblok H7 (45 mcg) Unadjuvanted (N=84)
Injection Site Pain (General disorders) | 53 (66) | 51 (60) | 7 (8)
Malaise (General disorders) | 33 (40) | 30 (33) | 15 (16)
Upper Respiratory Tract Infection (Infections and infestations) | 9 (9) | 9 (10) | 5 (5)
Myalgia (Musculoskeletal and connective tissue disorders) | 32 (43) | 37 (41) | 11 (13)
Headache (Nervous system disorders) | 36 (44) | 33 (41) | 12 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.

DOCUMENTS (2):
  • Study Protocol (2022-09-14): https://cdn.clinicaltrials.gov/large-docs/05/NCT05608005/Prot_000.pdf
  • Statistical Analysis Plan (2022-05-27): https://cdn.clinicaltrials.gov/large-docs/05/NCT05608005/SAP_001.pdf